CLINICAL TRIAL: NCT00587730
Title: Attenuation Corrected Cardiac SPECT Using the GE Hawkeye Camera System
Acronym: Hawkeye
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Recruiting or enrolling participants has halted prematurely and will not resume.
Sponsor: Mayo Clinic (Other)
Responsible Party: Todd D. Miller, MD/Professor of Medicine, Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1042-01
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Cardiac Disease
Keywords: heart disease; cardiac disease; chest pain; myocardial infarction; heart attack
MeSH Terms: conditions — Heart Diseases; Chest Pain; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Clinical SPECT (Active Comparator): GE Hawkeye Attenuation Correction Camera is being compared to the approved clinical use SPECT camera.
  Interventions: Device: GE Attenuation Corrected Hawkeye Camera

INTERVENTIONS:
Device: GE Attenuation Corrected Hawkeye Camera — GE Hawkeye AC system and 360˚ camera orbit

SUMMARY:
The accuracy of stress single photon emission computed tomography (SPECT) is limited by imaging artifacts, many of which are caused by soft tissue attenuation. A recent multicenter study performed by our laboratory comparing 7 commercially available attenuation correction (AC) camera systems in a cardiac phantom showed the best performance with the GE Hawkeye (a hybrid gamma camera-CT scanner) and the University of Michigan M-step (unique feature a camera orbit of 360˚ versus the usual 180˚) systems. In this study we will combine the strengths of these two systems (GE Hawkeye AC system and 360˚ camera orbit) to test the accuracy of this imaging system in a population of 400 consecutive patients undergoing clinically indicated stress SPECT. These patients will undergo SPECT imaging both with conventional methodology and the GE Hawkeye system. The conventional study will be interpreted and reported in the usual clinical fashion. The GE Hawkeye images will be interpreted independently by 2 observers blinded to the results of conventional imaging and will not be reported clinically. The primary study hypothesis is that AC will substantially reduce attenuation artifacts (mild fixed defects) without reducing the accuracy of either normal studies or myocardial infarction (MI). Clinical data and noninvasive test results (history of MI, electrocardiogram, and gated wall motion) will be used to distinguish defects which represent attenuation (false-positive) versus those due to MI (true-positive).

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to the Charlton Nuclear Cardiology Laboratory for stress Tc-99m sestamibi SPECT

Exclusion criteria:

* Prior PTCA or CABG
* Left bundle branch block (LBBB) or paced ventricular rhythm
* Clinically significant valvular heart disease
* Hypertrophic or idiopathic dilated cardiomyopathy
* Atrial fibrillation or frequent atrial or ventricular ectopy (defined as >20% ectopic beats
* History of MI
* ECG evidence of MI
* Chest circumference >55 inches

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 608 (Actual)
Dates: Start 2001-07; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
The overall comparisons of the agreement between conventional SPECT imaging and the GE Hawkeye system will be completed using McNemar's test. | Measured/Compared at time of each scan.

SECONDARY OUTCOMES:
Comparisons of categorical factors between the 2 tests will also be completed using McNemar's test, continuous factors will be completed using a paired t-test if the differences are normally distributed. | Measured/Compared at time of study

CONTACTS AND LOCATIONS:
Overall Officials: Todd D Miller, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States